CLINICAL TRIAL: NCT00861458
Title: A Phase 1, Open-Label, Randomized, 3-Way Crossover Study In Healthy Subjects To Estimate The Pharmacokinetics Of PF-00868554 Administered As 3x250mg Oral Tablets (Wet Granulate, 3x250mg Oral Tablets (Dry Granulate) And 750mg Solution Under Fed State
Brief Title: Bioavailability Study Of PF-00868554 Administered As 3x250mg Oral Tablets (Wet Granulate, 3x250mg Oral Tablets (Dry Granulate) And 750mg Solution Under Fed State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A8121010
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-00868554 (Experimental)
  Interventions: Drug: Pharmacokinetics

INTERVENTIONS:
Drug: Pharmacokinetics — Single dose of 750 mg PF-00868554 as a solution and tablets.
  Other Names: pharmacokintics

SUMMARY:
This study will test two different formulations. The results will be used to select formulation for phase 3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.

Exclusion Criteria:

* Standard for healthy volunteers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
AUC inf, Cmax | 2 days

SECONDARY OUTCOMES:
Adverse events | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121010&StudyName=Bioavailability%20Study%20Of%20PF-00868554%20Administered%20As%203x250mg%20Oral%20Tablets%20%28Wet%20Granulate%2C%203x250mg%20Oral%20Tablets%20%28Dry%20Granulate%29%20And%207